CLINICAL TRIAL: NCT04497064
Title: Breakfast Knowledge, Beliefs, and Habits of Exercising Adults
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Ohio University
Other Study IDs: 19-E-364
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Nutrition
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athlete: those who identified as participating in athletic competitions at DI, intramural, club or competitive levels
  Interventions: Other: survey
- non-athletes: those who did not identify as participating in athletic competitions at DI, intramural, club or competitive levels
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — survey asking questions regarding breakfast habits and composition, sports nutrition knowledge and exercise habits

SUMMARY:
This study is being done to determine typical breakfast consumption habits in various populations of exercisers. Participants will be asked a series of questions pertaining to their participation in regular exercise, their current breakfast consumption, food preferences, meal timing, and general knowledge of sports nutrition and pre-exercise breakfast consumption.

DETAILED DESCRIPTION:
Participants will complete a one-time survey regarding breakfast habits and beliefs and sports nutrition knowledge, as well as the type, frequency, and intensity of exercise engaged in on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* regular exerciser

Exclusion Criteria:

* younger than 18 years old
* do not regularly exercise

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: anyone with a valid Ohio University email address or who saw the advertisement on social media who was older than 18 and participates in structured exercise
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
breakfast composition | Day 1
  Questions asked include typical composition of breakfast, such as Meat, Plant-based protein (beans, lentils, peas), Nuts or seeds, Cheese, Eggs, Yogurt or dairy, Bread, Starchy vegetables, Non-starchy vegetables, Grains, Fruit/fruit juice, or Protein/meal replacement bars
breakfast habits | Day 1
  questions regarding typical breakfast consumption habits
breakfast beliefs | Day 1
  questions regarding how individuals felt about eating breakfast
sports nutrition knowledge | Day 1
  questions from the 49-SNKI to assess sports nutrition knowledge
exercise habits | Day 1
  questions on frequency, duration and intensity of typical exercise sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
upon request